CLINICAL TRIAL: NCT04561687
Title: Comparison of Montelukast and Azelastine in Treatment of Moderate to Severe Allergic Rhinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasrin Mortazavi Far, Principal investigator, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-01-49-21547
Record Dates: First submitted 2020-09-11; First posted 2020-09-24 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — montelukast; azelastine; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Azelastine and Nasal Budesonide (Active Comparator): Spray nasal Azelastine 1puff daily for 6-12years old patients and 2puff for older
  Interventions: Drug: Azelastine; Drug: Budesonide
- Montelukast and Nasal budesonide (Active Comparator): Montelukast 5mg 6-14years old and 10mg for older
  Interventions: Drug: Montelukast; Drug: Budesonide
- Nasal Budesonide and Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Budesonide; Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — Montelukast and nasal budesonide
  Arms: Montelukast and Nasal budesonide
Drug: Azelastine — Azelastine and nasal budesonide
  Arms: Azelastine and Nasal Budesonide
Drug: Budesonide — To all groups
Drug: Placebo — Placebo and nasal budesonide
  Arms: Nasal Budesonide and Placebo

SUMMARY:
Comparison of Montelukast and Azelastine In treatment of Allergic Rhinitis Allergic intent is one of the most common diseases of the respiratory system that has a devastating effect on the quality of life. The importance of studying this disease can be seen from the high prevalence of this diseas. In addition to the high prevalence, due to the reducing effect of this disease on the economy and academic performance of patients, a great burden is imposed by this disease on the country's health care system.Also finding the best treatment of allergic can help to control of Asthma if exists concurrently.

Inflammation of the nasal mucosa following the release of IgE can be shown as symptoms of runny nose, sneezing, nasal congestion.Many studies have been done in the field of allergic rhinitis to increase the cost-effectiveness of treatment of this complication. Among the treatments for this disease is the use of antihistamine nasal sprays such as Azelastine. Combination therapies such as combining Mometason furoate or fluticasone with Azelastine or Montelukast can also be mentioned. However, there is still a long way to go to find the best drug combination to reduce the economic and human costs to the global health system. Due to the high prevalence of allergic diseases such as allergic rhinitis, finding the best treatment or management of such diseases plays an important role in improving the quality of life and reducing the economic burden on society.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-50years
* Moderate to severe allergic rhinitis

Exclusion Criteria:

* Under any treatment

  * Drug sensitivity

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Sino-Nasal Outcome Test scores (SNOT-22) | Baseline,month1,month3
  Change in Sino-Nasal Outcome Test scores (SNOT-22) scores pre- and post-treatment. The Sino-Nasal Outcome Test asks subjects to rate how "bad" their rhinosinusitis by using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be.

CONTACTS AND LOCATIONS:
Overall Officials: Nasrin Mortazavi, Principal Investigator — Shiraz University of Medical Science
Locations (1):
- Shiraz University of Medical Science, Shiraz, Iran